CLINICAL TRIAL: NCT07252050
Title: Ruxolitinib-Enhanced Conditioning for Pediatric and Young Adult Patients With Symptomatic Sickle Cell Disease Undergoing Haploidentical Hematopoietic Cell Transplantation
Brief Title: Ruxolitinib-Enhanced Haplo HCT for Children and Young Adults With Sickle Cell Disease
Acronym: RUX-HAPLO
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Healthcare of Atlanta (Other); Emory University (Other); Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Laura McLaughlin, Lead Principal Investigator/Study Chair, University of Colorado, Denver
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-0735
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease; Hematopoetic Stem Cell Transplant; Haploidentical Hematopoietic Stem Cell Transplant; Haploidentical Stem Cell Transplantation; Graft Failure
Keywords: Sickle cell disease; Hematopoietic cell transplant; Ruxolitinib; Pediatric; Young Adult; Haplo
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ruxolitinib-Enhanced RIC (Experimental): Pediatric and young adult participants who are undergoing haplo HCT for SCD will receive RIC with fludarabine, cyclophosphamide, thiotepa, ATG and low-dose TBI along with ruxolitinib. Ruxolitinib will continue post-HCT in addition to post-transplant cyclophosphamide and sirolimus or a calcineurin inhibitor for GVHD prophylaxis.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — All participants will receive ruxolitinib beginning during conditioning in addition to conventional RIC and GVHD prophylaxis.
  Other Names: Jakafi

SUMMARY:
This trial will determine whether adding ruxolitinib to a reduced intensity conditioning (RIC) regimen reduces the rate of graft failure following haploidentical (haplo) hematopoietic cell transplant (HCT) for children and young adults with sickle cell disease (SCD).

This study will enroll and treat up to 24 participants. Recruitment is expected to last for about 2 years and participants will be followed for an additional 2 years post-HCT.

DETAILED DESCRIPTION:
While haplo HCT following a RIC regimen cures most patients with SCD, graft failure (GF) can occur and result in return of SCD. GF occurs more often in pediatric SCD patients and can be associated with significant morbidity and/or mortality. Development of strategies which reduce the risk of GF is needed to further improve haplo HCT outcomes for SCD, particularly in pediatric patients. This trial hopes to demonstrate that addition of ruxolitinib to a RIC regimen will reduce the incidence of GF without increasing conditioning-related toxicities.

The RUX-HAPLO study is a Phase 1/2 single-arm, multi-center, open-label trial for pediatric and young adult patients undergoing haplo HCT for SCD. The study will enroll up to 24 participants over approximately 2 years. All participants will receive cytoreduction with hydroxyurea (HU) for at least 60 days (Day -70 to Day -10) prior to the start of conditioning. All participants will then receive a RIC regimen consisting of cyclophosphamide, fludarabine, thiotepa, ATG and TBI beginning on Day -9. Ruxolitinib will begin during conditioning and will continue post-HCT. Participants will also receive GVHD prophylaxis with post-transplant cyclophosphamide, in addition to sirolimus or a calcineurin inhibitor.

The primary objective is to estimate 1-year event-free survival (EFS) with primary or secondary GF or death counting as events for this endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with any genotypic form of SCD aged 12 - 45 years at enrollment with ≥1 of the following:

   1. History of stroke and/or vasculopathy, including evidence of asymptomatic cerebrovascular disease for pediatric patients.
   2. Recurrent moderate-severe acute chest syndrome (ACS)
   3. Recurrent vaso-occlusive pain episodes requiring parenteral analgesia despite the institution of supportive care.
   4. Need for chronic transfusion therapy to prevent vaso-occlusive complications (i.e. pain, stroke, and ACS).
   5. For adult patients, an echocardiographic finding of tricuspid valve regurgitant jet velocity (TRJV) ≥ 2.7 m/sec.
2. Participants must have an HLA haploidentical first degree relative (parent, sibling, or half sibling) who is willing and able to donate bone marrow.
3. Participants must meet institutional eligibility criteria for HCT.

Exclusion Criteria:

1. Presence of an HLA-matched sibling who is willing and able to donate bone marrow.
2. Uncontrolled infection, evidence of active TB, Hepatitis B or C infection, or HIV seropositivity or infection.
3. Previous HCT or solid organ transplant.
4. CNS revascularization procedure, myocardial infarction, pulmonary embolus or deep vein thrombosis in the past 6 months.
5. Use of medications which significantly interfere with ruxolitinib metabolism.
6. Known hypersensitivity or severe reaction to ruxolitinib or any component of the conditioning regimen or its excipients.
7. Inability to swallow and retain oral medication (use of nasogastric or gastrostomy tube permitted).
8. History of malignancy except resected basal cell carcinoma or treated carcinoma in-situ.
9. Participation in another clinical trial involving an investigational or off-label use of a drug or device in the past 3 months.
10. Currently pregnant or breast feeding.
11. Clinically significant, uncontrolled autoimmune disease.
12. High-titer anti-donor specific HLA antibodies (without review and approval by Study Chair).
13. Participant (or guardian) inability or unwillingness to comply with the dose schedule and study evaluations, comprehend or sign informed consent and utilize a highly effective method of contraception (for participants of child-bearing potential).
14. Any condition that would, in the investigator's judgment, interfere with full participation in the study, pose a significant risk to the subject, or interfere with interpretation of study data.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-11-19 (Estimated); Study Completion 2029-11-19 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | 1 year post-HCT
  Event Free Survival (EFS) is defined as survival without a qualifying event (primary or secondary GF, second HCT or death).

SECONDARY OUTCOMES:
Overall Survival | 1 and 2 years post-HCT
  Overall survival will be described at 1 and 2 years post-HCT including death from any cause after HCT.
Event Free Survival | 2 years post-HCT
  Event Free Survival (EFS) is defined as survival without a qualifying event (primary or secondary GF, second transplant or death).
Neutrophil Recovery | Up to Day 60 post-HCT
  The time to neutrophil recovery, in days, will be reported. Neutrophil recovery is defined as the first of 3 measurements on different days when the absolute neutrophil count is ≥500/μL after nadir.
Platelet Recovery | Up to Day 180 post-HCT
  The time to platelet recovery, in days, will be reported. Platelet recovery is defined as the first day the platelet count is ≥50,000/μL of blood, without a transfusion in the preceding 7 days with the exception of a platelet transfusion specifically to achieve a platelet threshold to allow an elective invasive procedure.
Acute GVHD | Up to Day +100 post-HCT
  Incidence of overall and severe (Grade 3-4) acute GVHD (based on MAGIC criteria) will be estimated at until Day 100 post-HCT.
Chronic GVHD | 6 months to 2 years post-HCT
  Incidence of overall and severe chronic GVHD (according to the NIH consensus criteria) will be estimated at 6 months, 1 year, 18 months and 2 years post-HCT.
Donor hematopoietic chimerism | Day 28 to 2 years post-HCT
  Characterization of donor chimerism in peripheral blood for lymphoid and myeloid fractions will be performed at day 28, 60, 100, and 180 and 1 and 2 years post-HCT.
Primary Graft Failure | Day 42 post-HCT
  The incidence of primary graft failure (GF) by day 42 post-HCT will be estimated. Primary GF is defined as never achieving ≥ 5% donor whole blood or myeloid chimerism. Second infusion of stem cells is also considered indicative of primary GF.
Secondary Graft Failure | Up to 2 years post-HCT
  The incidence of secondary graft failure (GF) by 2 years post-HCT will be estimated. Secondary GF is defined as < 5% donor whole blood or myeloid chimerism beyond day +42 post-HCT in participants with prior documentation of hematopoietic recovery with > 5% donor cells by day +42 post-HCT. Second infusion of stem cells beyond Day +42 is also considered indicative of secondary GF.
Hepatic VOD/SOS | Up to 2 years post-HCT
  The incidence of hepatic veno-occlusive disease (VOD)/sinusoidal obstruction by 2 years post-HCT will be estimated.
IPS | Up to 2 years post-HCT
  The incidence of idiopathic pneumonia syndrome (IPS) by 2 years post-HCT will be estimated.
CNS Toxicity | Up to 2 years post-HCT
  The incidence of CNS toxicity, defined as seizures, intracranial hemorrhage (ICH), posterior reversible encephalopathy syndrome (PRES) or reversible posterior leukoencephalopathy syndrome (RPLS) will be estimated.
Significant infections | Up to 2 years post-HCT
  The incidence of cytomegalovirus (CMV) infection, adenovirus infection, Epstein-Barr Virus (EBV) post-transplant lymphoproliferative disease (PTLD), or other clinically significant viral reactivations, invasive fungal infections and bacterial sepsis will be estimated.
Prolonged Immunosuppressive Therapy | Up to 2 years post-HCT
  The proportion of participants receiving immunosuppressive therapy beyond 1 year post-HCT because of GVHD or concerns about graft rejection will be determined.
SCD-related Complications | Up to 2 years post-HCT
  SCD-related complications at 6 months, 1 and 2 years post-HCT will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Laura McLaughlin, MD, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Manning Family Children's, New Orleans, Louisiana
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No